CLINICAL TRIAL: NCT01522781
Title: 10 Year Outcome of Total Knee Replacement (TKR) Using Sigma Prosthesis
Status: Completed | Type: Observational
Sponsor: NHS Fife (Other Government)
Collaborators: DePuy International (Industry)
Responsible Party: Principal Investigator, Ivan Brenkel, Consultant Orthopaedic Surgeon. Lead investigator, NHS Fife
Other Study IDs: IIS2010001
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to obtain a prospective database which will allow analysis of total knee outcomes.

DETAILED DESCRIPTION:
A prospective database was set up in October 1998. Patient details are collected pre-operatively, intra-operatively and immediately post operatively. Patients are then followed up in a dedicated knee clinic at 6 months, 18 months, 3 years and 5 years. Data such as SF12 and the American knee society score has been done at each visit.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing total knee replacement in Fife

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing total knee replacement in Fife
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 1998-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Clinical outcome of the Sigma knee at 10 years | 10 years
  Patient satisfaction scores SF 12 and Oxford American Knee society score

SECONDARY OUTCOMES:
Radiographic outcomes at 10 years | 10 years
  looking for failure by identitying lucent lines and osteolysis

CONTACTS AND LOCATIONS:
Locations (1):
- Fife Health Board, Kirkcaldy, Fife, United Kingdom